CLINICAL TRIAL: NCT03281525
Title: Sleep Quality: Comparison Between Patients With VAD and Patients That Underwent Heart Transplant, an Observational Study
Brief Title: Sleep Quality Underwent Heart Transplant, an Observational Study
Acronym: SQ_Heart
Status: Completed | Type: Observational
Sponsor: University of Padova (Other)
Responsible Party: Sponsor
Other Study IDs: SQ_Heart2017
Record Dates: First submitted 2017-09-05; First posted 2017-09-13 (Actual); Last update posted 2020-12-04 (Actual); Status verified 2020-12

CONDITIONS: Ventricular Dysfunction
Keywords: cardiotransplant
MeSH Terms: conditions — Ventricular Dysfunction

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The SQ_Heart has been designed as an observational study that evaluates the difference in sleep quality between 11 patients with VAD (Ventricular Assisted Device) and 98 Cardiotransplant patients.

DETAILED DESCRIPTION:
The Primary objective of the SQ_Heart study is to evaluate the significant difference in sleep quality between patients with VAD (Ventricular Assisted Device) and cardiotransplant patients, using the Pittsburgh scale Sleep Quality Index (PSQI), with a cut-off of > 5 for poor sleepers.

Patients, to be enrolled, must provide:

* Age ≥ 18 and < 90;
* Cardiotransplant patients, with VAD or non;
* patients with VAD.
* subjects able to sign informed consent.

All the patients will have to complete some questionnaires:

* questionnaire about the diagnosis of pathology and lifestyle;
* questionnaire about the perceived quality of sleep through the use of Pittsburgh Sleep Quality (PSQI);
* questionnaire about the perceived quality of life (Euro Quality of Life 5D-5L).

Questionnaires are necessary for the data collection for the study.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 and < 90;
* Cardiotransplant patients, with VAD (Ventricular Assisted Device) or non;
* patients with VAD ;
* subjects able to sign informed consent.

Exclusion Criteria:

* Age < 18;
* subjects don't sign informed consent;
* hospitalization for more than 30 days before compilation in intensive care unit.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cardiotransplant patients with VAD (Ventricular Assisted Device) or non; Patients with VAD
Sampling Method: Probability Sample
Enrollment: 176 (Actual)
Dates: Start 2017-04-11 (Actual); Primary Completion 2017-09-30 (Actual); Study Completion 2017-09-30 (Actual)

PRIMARY OUTCOMES:
Sleep Quality Index | up 30 days
  sleep quality

CONTACTS AND LOCATIONS:
Locations (1):
- Azienda Ospedaliera di Padova, Padua, Italy